CLINICAL TRIAL: NCT00349817
Title: Genetics Education: Preparing Physicians for the Future
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: University of Toronto
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2006-07-10 (Estimated); Status verified 2006-07

CONDITIONS: Primary Care Genetics; Hereditary Colorectal Cancer

INTERVENTIONS:
Behavioral: web-based learning, didactic lecture and role-play

SUMMARY:
This study examines the best way to teach genetics to family medicine residents. First year family medicine residents at the University of Toronto will be taught basic clinical genetics as well as a specific disease in genetics via 3 different educational methods. All participants will undergo an oral examination and written knowledge test 3 months after this education. Results between groups will be compared, and the best way to teach genetics to residents determined.

DETAILED DESCRIPTION:
An educational module will be prepared by the investigators outlining important genetic fundamentals and hereditary colorectal cancer. Sixty four family medicine resident participants will take part in this study. Participants will be divided into 4 groups. Group 1 will be the control and receive no education. Group 2 will be given access to the self-study web-based educational module to do on their own time. Group 3 will be given a lecture on the material using the educational module, followed by a discussion. Group 4 will also be given this lecture and discussion, followed by an interactive standardized patient role-play experience.

Three months later, all participants will complete an simulated oral examination, an written knowledge test and an attitude survey. By comparing the results between the 4 groups, the best way to teach genetics will be determined. This template can then be used to develop a curriculum for teaching clinical genetics to family medicine residents.

ELIGIBILITY:
Inclusion Criteria:

* all first year family medicine residents in the Department of Family and Community Medicine at the University of Toronto

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 2005-10; Study Completion 2007-01

PRIMARY OUTCOMES:
knowledge in approach to family medicine genetics
attitude towards family medicine genetics and genetic testing
skill in discussing these issues with patients

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Telner, MD, MED, CCFP, Principal Investigator — Department of Family and Community Medicine, University of Toronto
Locations (1):
- Deanna Telner, Toronto, Ontario, Canada